CLINICAL TRIAL: NCT01074307
Title: Prospective, Open-labeled Trial in Patients With Systolic Heart Failure to Evaluate Bisoprolol Treatment for the Effects on Surrogate Markers of Heart Failure in Korea (PRISM)
Brief Title: A Prospective, Open-labeled, Multi-centric Trial in Subjects With Systolic Heart Failure to Evaluate Bisoprolol Treatment for the Effects on Surrogate Markers of Heart Failure in Korea
Acronym: PRISM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMD 084000-608
Record Dates: First submitted 2010-02-22; First posted 2010-02-24 (Estimated); Results first posted 2014-02-14 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-01

CONDITIONS: Heart Failure, Congestive
Keywords: Systolic heart failure; Bisoprolol; Concor; Echocardiogram
MeSH Terms: conditions — Heart Failure; Heart Failure, Systolic | interventions — Bisoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Dose Bisoprolol (Experimental)
  Interventions: Drug: Low Dose Bisoprolol
- High Dose Bisoprolol (Experimental)
  Interventions: Drug: High Dose Bisoprolol

INTERVENTIONS:
Drug: Low Dose Bisoprolol — Bisoprolol tablet (Concor) will be administered orally at a starting dose of 1.25 milligram (mg) once daily for 2 weeks. The dose will be further escalated from 1.25 mg to 2.5 mg once daily after 2 weeks and will be administered up to 26 weeks, only if the previous administered dose is well tolerated. If the subject could not tolerate the increased dose, then the last tolerated dose will be maintained up to 26 weeks.
  Other Names: Concor
  Arms: Low Dose Bisoprolol
Drug: High Dose Bisoprolol — Bisoprolol tablet (Concor) will be administered orally at a starting dose of 3.75 mg once daily for 2 weeks. The dose will be subsequently increased to 5 mg, 7.5 mg, or 10 mg once daily every two weeks and will be administered up to 26 weeks, only if the previous administered dose is well tolerated. If the subject could not tolerate the increased dose, then the last tolerated dose will be maintained up to 26 weeks.
  Other Names: Concor
  Arms: High Dose Bisoprolol

SUMMARY:
This is a prospective, open-labeled, multi-centric trial to evaluate the effect of bisoprolol (between low dose and high dose) on surrogate markers of heart failure in Korea.

DETAILED DESCRIPTION:
Subjects with systolic congestive heart failure (CHF) will be enrolled in this study after proper evaluation of NT-proBNP, global assessment of CHF, 6-minute walking test and improvement score of New York Heart Association (NYHA) and echocardiogram (left ventricular chamber size and ejection fraction [LVEF]). Each subject will be orally administered bisoprolol for 6 months starting at 1.25 mg at the Week 0 and titrated up to 10 mg during the 6 month period if the persistent standing systolic blood pressure (SBP) is greater than (>) 90 millimeter of mercury (mm Hg) and there is no symptom of hypotension at the current dose medication (syncope, loss of consciousness, dizziness when standing up).

OBJECTIVES

Primary objective:

• To evaluate the effect of bisoprolol (between low dose and high dose) on surrogate markers of heart failure in Korea

Secondary objectives:

* To evaluate bisoprolol for the effects on clinical improvement of heart failure in Korea:

  1. New York Heart Association (NYHA),
  2. 6-minutes walking test
  3. Echocardiogram (left ventricular chamber size and LVEF)
* Hospitalization due to heart failure
* To evaluate the safety and tolerability of bisoprolol
* Global assessment of CHF

ELIGIBILITY:
Inclusion Criteria:

* Subjects with heart failure and at the age of 18 (inclusive) to 80 (exclusive)
* Subjects with NYHA Class II-IV with dyspnea
* Subjects with left ventricular ejection fraction (LVEF) of 40 percent or below on the echocardiogram
* Eligible subjects who meet the criteria, are capable of participating in the study, and provide written informed consent to study participation after receiving a clear explanation about the study objective and nature

Exclusion Criteria:

* A subject who cannot understand or does not agree to the study contents
* Subjects with conduction defect of 2nd degree or above atrioventricular block
* Subjects with heart rate less than (<) 60 beats at rest
* Subjects with systolic blood pressure < 100 mm Hg at rest
* Subjects with renal failure (serum creatinine > 2.0 milligram per deciliter [mg/dL])
* Subjects with unrecovered pulmonary edema
* Subjects with history of myocardial infarction or stroke within 3 months
* Subjects with history of coronary intervention or coronary bypass within 6 months
* Subjects with heart failure due to mitral valve without valve replacement or aortic valvular disease (excluding moderate or less severe mitral insufficiency secondary to left ventricular expansion)
* Subjects with history of valve replacement within the past 6 months
* Subjects with history or scheduled heart transplantation
* Subjects with reversible obstructive pulmonary disease
* Subjects with other cases where beta blockers are contraindicated
* Any surgical or internal disease that may put the subject at a higher risk due to study participation or may interfere with the subjects compliance to study requirements or completion of the study, based on the judgment of the Investigator
* A subject with history of non-compliance to drug prescriptions or who is not willing to comply with the protocol
* Subjects with a history of treated or untreated malignant tumor within the past 5 years
* Pregnant or lactating women
* Subjects with heart failure due to acute myocarditis
* Subjects with continuous ventricular tachycardia with history of syncope within 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2009-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Ltd.
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose Bisoprolol: Bisoprolol tablet (Concor) administered orally at a starting dose of 1.25 milligram (mg) once daily for 2 weeks. The dose was further escalated from 1.25 mg to 2.5 mg once daily after 2 weeks and was administered up to 26 weeks, only if the previous administered dose was well tolerated. If the participant didn't tolerate the increased dose, then the last tolerated dose was maintained up to 26 weeks.
- High Dose Bisoprolol: Bisoprolol tablet (Concor) administered orally at a starting dose of 3.75 mg once daily for 2 weeks. The dose was subsequently increased to 5 mg, 7.5 mg, or 10 mg once daily every two weeks and was administered up to 26 weeks, only if the previous administered dose was well tolerated. If the participant didn't tolerate the increased dose, then the last tolerated dose was maintained up to 26 weeks.
Period: Overall Study
Arm/Group | Low Dose Bisoprolol | High Dose Bisoprolol
Started | 66 | 114
Completed | 44 | 102
Not Completed | 22 | 12
Not completed — No primary endpoint evaluation | 14 | 6
Not completed — Exclusion criterion | 0 | 1
Not completed — Protocol Violation | 8 | 5

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) population included all the randomized participants who had at least one dose of the investigational product. Baseline data has been provided for 159 participants (ITT population).
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Bisoprolol | High Dose Bisoprolol | Total
Number analyzed (Participants) | 52 | 107 | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.88 (11.52) | 57.68 (12.28) | 59.38 (12.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 83 | 117
  Male | 18 | 24 | 42

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in N-terminal Pro B-type Natriuretic Peptide (NT-proBNP) at Week 26
Description: B-type natriuretic peptide (BNP) is a substance secreted from the ventricles or lower chambers of the heart in response to changes in pressure that occur when heart failure develops and worsens. The level of BNP in the blood increases when heart failure symptoms worsen, and decreases when the heart failure condition is stable. The BNP level in a person with heart failure is higher than in a person with normal heart function. The percent change of NT-pro BNP was calculated according to the formula: N-terminal pro B-type natriuretic peptide (NT-proBNP) reduction ratio = 100*(Baseline NT-proBNP - Week 26 NT-proBNP)/Baseline NT-proBNP.
Time Frame: Baseline and Week 26
Population: ITT population included all the randomized participants who had at least one dose of the investigational product. 'N' (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Low Dose Bisoprolol | High Dose Bisoprolol
Number analyzed (Participants) | 51 | 107
Percent change | 8.02 (113.78) | 9.50 (117.56)

2. Secondary Outcome: Percentage of Participants Classified as Class I to IV According to New York Heart Association (NYHA)
Description: New York Heart Association (NYHA) classification of heart failure: Class I: No limitation: ordinary physical exercise does not cause undue fatigue, dyspnea, or palpitations. Class II: Slight limitation of physical activity: comfortable at rest but ordinary activity results in fatigue, palpitations, or dyspnea. Class III: Marked limitation of physical activity: comfortable at rest but less than ordinary activity results in symptoms. Class IV: Unable to carry out any physical activity without discomfort: symptoms of heart failure are present even at rest with increased discomfort with any physical activity.
Time Frame: Baseline and Week 26
Population: ITT population included all the randomized participants who had at least one dose of the investigational product.
Measure: Number; unit: Percentage of participants
Arm/Group | Low Dose Bisoprolol | High Dose Bisoprolol
Number analyzed (Participants) | 52 | 107
Percentage of participants
  Baseline: Class II | 73.08 | 74.77
  Baseline: Class III | 25.00 | 24.30
  Baseline: Class IV | 1.92 | 0.93
  Week 26: Class I | 21.15 | 42.06
  Week 26: Class II | 69.23 | 54.21
  Week 26: Class III | 9.62 | 3.74

3. Secondary Outcome: Change From Baseline in 6-minute Walking Test (6-MWT) Distance at Week 26
Description: 6-minute Walking Test (6-MWT) distance was the distance that a participant could walk in 6 minutes. Participants were asked to perform the test at a pace that was comfortable to them, with as many breaks as they needed.
Time Frame: Baseline and Week 26
Population: ITT population included all the randomized participants who had at least one dose of the investigational product. 'N' (number of participants analyzed) signifies participants who were evaluable for this measure. 'n' signifies number of participants who were evaluable for specified categories at different time points.
Measure: Mean (Standard Deviation); unit: Meter
Arm/Group | Low Dose Bisoprolol | High Dose Bisoprolol
Number analyzed (Participants) | 52 | 103
Meter
  Baseline (n=52, 103) | 347.58 (123.35) | 368.11 (169.04)
  Change at Week 26 (n=47, 102) | 41.59 (103.45) | 28.45 (161.66)

4. Secondary Outcome: Change From Baseline in Echocardiographic Left Ventricular Ejection Fraction (LVEF) at Week 26
Description: LVEF was defined as the fraction of blood (in percent) pumped out of the heart's left ventricular chamber with each heart beat and it is used to measure the cardiac output for the heart.
Time Frame: Baseline and Week 26
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent LVEF
Arm/Group | Low Dose Bisoprolol | High Dose Bisoprolol
Number analyzed (Participants) | 52 | 106
Percent LVEF
  Baseline (n=52, 106) | 28.68 (7.47) | 27.61 (6.72)
  Change at Week 26 (n=50, 106) | 8.83 (9.47) | 14.22 (11.81)

5. Secondary Outcome: Change From Baseline in Echocardiographic Left Ventricular Size at Week 26
Description: Left ventricle size was measured as systolic and diastolic Left Ventricular Internal Dimension (LVID). Diastolic dimension was measured of the left ventricle at the level of the chordae tendineae. The systolic dimension was measured as the smallest dimension between the left septal endocardium and the posterior wall endocardium during systole, whether or not the two walls were exactly apposed.
Time Frame: Baseline and Week 26
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Milliliter LVID
Arm/Group | Low Dose Bisoprolol | High Dose Bisoprolol
Number analyzed (Participants) | 52 | 106
Milliliter LVID
  Baseline: Systolic LVID (n=51, 104) | 54.25 (8.80) | 54.69 (8.95)
  Change at Week 26: Systolic LVID (n=47, 102) | 5.46 (7.25) | 9.84 (9.32)
  Baseline: Diastolic LVID (n=52, 106) | 64.28 (7.99) | 63.40 (7.87)
  Change at Week 26: Diastolic LVID (n=50, 106) | 3.12 (4.37) | 5.49 (8.45)

6. Secondary Outcome: Number of Participants Who Were Re-hospitalized Due to Heart Failure and Who Died Due to Cardiovascular Disorder
Time Frame: Baseline up to Week 26
Population: ITT population included all the randomized participants who had at least one dose of the investigational product.
Measure: Number; unit: Participants
Arm/Group | Low Dose Bisoprolol | High Dose Bisoprolol
Number analyzed (Participants) | 52 | 107
Participants
  Re-hospitalization due to heart failure | 3 | 3
  Death due to cardiovascular disorder | 0 | 0

7. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to baseline during a clinical study with an Investigational Medicinal Product (IMP), regardless of causal relationship and even if no IMP has been administered.
Time Frame: Baseline up to Week 26
Population: Safety analysis population included all the randomized participants who had at least one dose of the investigational product had post-dose safety data confirmed at least once by the Investigator.
Measure: Number; unit: Participants
Arm/Group | Low Dose Bisoprolol | High Dose Bisoprolol
Number analyzed (Participants) | 66 | 114
Participants | 45 | 73

8. Secondary Outcome: Mean Change From Baseline in Global Assessment of Congestive Heart Failure (CHF) Score at Week 26
Description: Global assessment of CHF: The Investigator defined, graded, and recorded the participant's symptoms and signs by using a 6-point CHF scale ranging from 0 (unassessable), 1 (worsened), 2 (no change), 3 (mildly improved), 4 (moderately improved) and 5 (markedly improved).
Time Frame: Baseline and Week 26
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Low Dose Bisoprolol | High Dose Bisoprolol
Number analyzed (Participants) | 52 | 106
Units on a scale
  Baseline (n=52, 106) | 2.52 (1.02) | 2.71 (0.92)
  Change at Week 26 (n=51, 106) | 0.45 (1.27) | 0.69 (1.41)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 26
Description: An AE is defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to baseline during a clinical study with an IMP, regardless of causal relationship and even if no IMP has been administered.
Arm/Group | Low Dose Bisoprolol | High Dose Bisoprolol
Serious Adverse Events (participants affected / at risk) | 16/66 | 9/114
Other Adverse Events (participants affected / at risk) | 45/66 | 71/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose Bisoprolol (N=66) | High Dose Bisoprolol (N=114)
Cardiac failure (Cardiac disorders) | 1 | 2
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 1 | 2
Chest discomfort (General disorders) | 1 | 0
Chest Pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Sudden cardiac death (General disorders) | 2 | 1
Diabetic foot (Metabolism and nutrition disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0
Insomnia (Nervous system disorders) | 1 | 0
Flank pain (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose Bisoprolol (N=66) | High Dose Bisoprolol (N=114)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 11
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Cardiac failure (Cardiac disorders) | 1 | 4
Hypotension (Vascular disorders) | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 4
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Dizziness (Nervous system disorders) | 10 | 15
Insomnia (Psychiatric disorders) | 3 | 1
Asthenia (General disorders) | 2 | 6
Chest discomfort (General disorders) | 6 | 3
Oedema (General disorders) | 0 | 9
Oedema peripheral (General disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator commits him/her to forward to sponsor all papers, manuscripts or conference abstracts intended for publication or presentation that contain data or results generated in connection with the study. Papers and abstracts must be available at sponsor's site in time before the planned submission date to allow for review and comments. Submission for publication need expressed written permission from the sponsor. Any publication should follow publication policy as described in protocol.